CLINICAL TRIAL: NCT05577533
Title: Digital Epidemiology Study on Brain Functioning in Children Aged 7 to 12 Years
Brief Title: Digital Epidemiology Study on Brain Functioning
Acronym: EPIDIA4Kids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: O-Kidia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-A00766-37; 2022-002949-17 (EudraCT Number)
Record Dates: First submitted 2022-09-16; First posted 2022-10-13 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-04

CONDITIONS: Child Development; Child Development Disorder
Keywords: Digital Epidemiology; Child; Neurodevelopment; Neurodevelopmental disorders; Mental disorders
MeSH Terms: conditions — Developmental Disabilities; Neurodevelopmental Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- O-Kidia battery (Other): A one-time visit will be performed in children aged 7 to 12 years old as follow :
  Children will be playing on a series of games with a touch screen tablet while video, EEGs and digit trajectories data will be collected from this mobile device
  1. Video recording of the participants during the tablet testing via the intrinsic camera - 30 min
  2. Assessments - Paper and tablet psychometric tests will be used during the administrations, 1h45
  3. Child health questionnaires - Questionnaires will be completed by children and parents during the visit, 20 min for each
  Interventions: Behavioral: O-Kidia game battery; Behavioral: O-Brain

INTERVENTIONS:
Behavioral: O-Kidia game battery — Children will be playing on a series of games with a touch screen tablet while video and digit trajectories data will be collected from this mobile device to analyze eye-, face-, sound-recognition.
Behavioral: O-Brain — Electrical recordings and measurements - A mobile EEG headset will be used during the visit - 30 min

SUMMARY:
Neurobiology has improved the integrative understanding of brain development. With digital technologies, digital (bio)markers would be relevant variables for a better understanding of the heterogeneity of cognitive and behavioral functioning in developing children.

However, the dominant statistical approach of group comparison tends to ignore intragroup variability. Applying high-dimensional data sets through multivariate methods and then combining their scores via predictive model learning algorithms would allow the identification of subtypes. Thus, EPIDIA4KIDS wants to understand the brain functioning of children aged 7 to 12 years old from heterogeneous data sources collected from a touchscreen tablet.

DETAILED DESCRIPTION:
The overall objective of the EPIDIA4KIDS study is to understand brain functioning in children aged 7 to 12 years from heterogeneous digital data collected with a touch tablet. The investigators want to develop a digital e-screening, similarly to a blood test result, for cognitive, emotional and behavioral performances in children from 7 to 12 years old, resulting from a multimodal and multi-stream analysis generated by an artificial intelligence algorithm.

The main aims are therefore to:

* Develop a normative base of cognitive, emotional and, behavioral performances with children aged 7 to 12 years old using our digital tool.
* Examine the validity of our e-assessment by comparing the generated results to those obtained with standard measures of convergent validity.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls
* Aged 7 to 12 years
* Fluent in the French language
* Agreement and signature of informed consent by the child
* Agreement and signature of informed consent by one of the legal representatives
* Estimated intelligence quotient > 85

Exclusion Criteria:

* No biological parent or legal guardian is able to give permission for the minor and agrees to participate in parental assessments
* Prematurity or other perinatal complications that required significant intervention
* History of neurological disorders, including seizure disorders, cerebral palsy, or other conditions requiring neurological or medical care :
* History of head injury:

  * Head trauma more than one year old with loss of consciousness >30 minutes, OR
  * Had to be hospitalized for head trauma, OR
  * Amnesia > 24 hours, OR
  * Confusion or loss of orientation >24 hours, OR
  * A brain scan revealed problems following a head injury, OR
  * Head trauma within the past year with loss of consciousness >10 minutes. Current or persistent major Axis I psychiatric disorder that may interfere with successful completion of the protocol (e.g., psychosis and bipolar disorder), or substance use disorder.

Current use of medications with significant effects on brain function or blood flow (e.g., antipsychotics, mood stabilizers); Attention Deficit Hyperactivity Disorder (ADHD) medications and Selective Serotonin Reuptake Inhibitors (SSRIs) are not excluded as the use of these medications is associated with certain neurodevelopmental disorders and assessment of these individuals will provide useful data to the community Not fluent in French (all youth materials are in French) Uncorrectable visual, hearing, or sensorimotor impairment, as the protocol items may not be valid.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 736 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Measure number of criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  Total errors, Number of errors in total, False responses
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Measure number of criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  False responses
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Measure number of criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  Number of responses other than omission
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Measure number of criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  Hits/Accuracy, Number of correct responses, Hits of correct responses
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Measure number of criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  Standard deviation of the 3 standard errors calculated for each task block
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Measure number of criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  Order of combination of responses
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Time criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of typically developing children when playing with the O-Kidia battery on a touchscreen tablet
  Hits of Reaction time (RT), Median of reaction times for correct responses, Hits RT SE Standard error of Hits RT, Hits RT block change
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Time criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of typically developing children when playing with the O-Kidia battery on a touchscreen tablet
  Slope of change in RT between blocks, Slope of change in RT standard errors between blocks
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Time criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of typically developing children when playing with the O-Kidia battery on a touchscreen tablet
  SE variability Standard deviation of the 3 standard errors calculated for each task block
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Time criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of typically developing children when playing with the O-Kidia battery on a touchscreen tablet
  Order of combination of responses by reaction time
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Eye-movement criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  - Eye-tracking associated with O-Kidia battery: Number of saccade (pro/anti-), Number of blinks
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Eye-movement for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  - Eye-tracking associated with O-Kidia battery: near-point convergence, Near-point contact point
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Eye-movement criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  - Eye-tracking associated with O-Kidia battery: amplitude, direction, direction interval,
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Time of eye-movement criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  - Eye-tracking associated with O-Kidia battery: reaction time, fixation, time interval
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Digit-movement criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  - Digit-tracking associated with O-Kidia battery : direction, cumulated distance, distance to the proper trajectory
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Time of digit-movement criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
  - Digit-tracking associated with O-Kidia battery : exploration time, time to the proper trajectory
Create a Normative Database for emotional, behavioral and cognitive performance | 24 months
  Velocity of digit-movement criteria for motor skills, emotions, cognition and behavior, and therefore a neurodevelopmental presentation of developing children when playing with the O-Kidia battery on a touchscreen tablet
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - Accuracy measures are :Total errors, Number of errors in total
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - False responses, Number of responses other than omission
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - Number of correct responses, Hits of correct responses
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - SE variability Standard deviation of the 3 standard errors calculated for each task block
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - Order of combination of responses
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - Reaction time (RT) median for correct responses, Hits RT SE Standard error of Hits RT, Hits RT block change
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - Slope of change in RT between blocks, Slope of change in RT standard errors between blocks
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : WISC-V subtests, including Verbal concept, Fluid Reasoning scale, Working Memory measures, Processing Speed abilities
  - SE variability Standard deviation of the 3 standard errors calculated for each task block, Order of combination of responses by reaction time
Convergence validity for the O-Kidia battery | 18 months
  Describe the subgroup and compare it to pattern of comorbidities : Event planification abilities, the Tower of London
  Determination of performance at the test of the Tower of London coupled with eye-tracking.
  * Tower of London: analysed variables are: Number of problems solved (maximum duration is one minute) Failure if three successive problems are unsolved Types of error : systematic rule violation, back-and-forth Percentage of problems solved with the execution (minimal) number of moves.
  * Hits/Accuracy Number of correct responses
  The higher score is the better outcome.
Convergence validity for the O-Kidia battery | 18 months
  Describe the subgroup and compare it to pattern of comorbidities : Event planification abilities, the Tower of London
  Time for the performance at the test of the Tower of London coupled with eye-tracking.
  * Duration for planification and execution
  * Reaction Time, Total errors
  * Hits RT Median of reaction times for correct responses, Hits RT SE Standard error of Hits RT
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Children Behavior Check List (short version, 32 items) 32 items rated on a 3-point Likert-type scale, ranging from "never" (0) to "very often" (3) for the anxiety scale. The higher score is the worse outcome.
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Children Behavior Check List (short version, 32 items) 32 items rated on a 3-point Likert-type scale, ranging from "never" (0) to "very often" (3) for the evitant/depression scale. The higher score is the worse outcome.
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Children Behavior Check List (short version, 32 items) 32 items rated on a 3-point Likert-type scale, ranging from "never" (0) to "very often" (3) for the social problem scale. The higher score is the worse outcome.
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Behavioral assessment of executive function scoring (BRIEF, 72 items)
  72 items rated on a 3-point Likert-type scale, ranging from "never" (1) to "often" (3).The clinical scale gives a well-rounded picture of the behavior of the child or adolescent being rated.
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : (Keith Conners-3, 108 items)
  -108-items rated on a 4-point Likert-type scale, ranging from "never" (0) to "often" (3) to give insight into ADHD assessment as well as comorbid disorders such as Oppositional Defiant Disorder and Conduct Disorder. The higher score is the worse outcome
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Autism Quotient List version scoring (10 items)
  -10-items rated on a 4-point Likert-type scale, ranging from "Strongly agree" (1) to "definitely disagree" (3). Only one point can be awarded for each question. Give 1 point for "Strongly agree" or "Definitely disagree " for questions 1, 5, 7, and 10. Award 1 point for "Strongly Disagree" or "Strongly Disagree" for each of questions 2, 3, 4, 6, 8 and 9. If the person scores 6 or higher, he or she probably has social difficulties requiring referral for a specialized diagnostic assessment.
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : QTAC scoring, coordination acquisition disorder (15 items)
  15-items rated on a 5-point Likert-type scale, ranging from "not alike" (1) to "extremyly alike disagree" (5). The higher the scores the higher coordination acquisition disorder is suspected.
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Inattention and Hyperactivity-Impulsivity components with the ADHD-Rating Scale (18 items)
  - Measure of number of criteria for inattention, hyperactivity-impulsivity and therefore clinical presentation of ADHD (Predominant Inattentive, Predominant Hyperactive-Impulsive, Combined )
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Inattention and Hyperactivity-Impulsivity components with the ADHD-Rating Scale (18 items)
  - ADHD Rating Scale: 9 inattention items and 9 hyperactivity-impulsivity items rated on a 0-3 scale (range 0-27), therefore the total score is on a 0-54 range. The higher the scores the higher the inattention and hyperactivity-impulsivity
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Perseverance
  - the Grit-Scale for Children (GSCA, 12 items), items rated on a 1-5 scale, therefore the total score is on a 0-60 range, then divided by 12. The maximum score on this scale is 5 (extremely gritty), and the lowest scale on this scale is 1 (not at all gritty).
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Motivation
  - the School Motivation Questionnaire (SMQ, 10 min), 30 items on a Five-point Likert-type scale, ranging from "never" (1) to "very often" (5). The SMQ maximum total score is 150 and the minimum is 30 with solid loading scores: Self-Determination (SD), Self-Efficacy (SE), Intrinsic Motivation (IM), and Grade Motivation (GM)
Convergence validity for the O-Kidia battery | 24 months
  Describe the subgroup and compare it to pattern of comorbidities : Sleep quality (Pittsburgh Sleep Quality Index, 11 items)
  - The PSQI consists of 11 self-report questions that combine to give 7 "components" of the overall score, with each component receiving a score from 0 to 3. In all cases, a score of 0 indicates no difficulty while a score of 3 indicates severe difficulty. The 7 components of the score are added together to give an overall score ranging from 0 to 21 points, with 0 indicating no difficulty and 21 indicating major difficulty. A global score is the addition of these 7 components.

SECONDARY OUTCOMES:
Description of participants' characteristics | 24 months
  Measure of demographics with age
Description of participants' characteristics | 24 months
  Measure of language spoken
Description of participants' characteristics | 24 months
  Measure of family structure, school, medical history with questionnaires
Description of participants' characteristics | 24 months
  Measure of manual laterality, Edinburgh handedness, short version, to indicate manual laterality from 4 items rated on a five-point Likert-type scale, ranging from "always right" to "always left", scoring from +100 to -100.
Description of participants' characteristics | 24 months
  Socioeconomic status as measure INSEE index
mobile EEG biomarkers | 24 months
  P300 wave amplitude and latency - Quantitative electroencephalography (qEEG) will be recorded during a resting state, Elicitation of evoked potentials (ERP) will use the O-Kidia battery to elicit components associated with attention, working memory, stress, or anxiety
mobile EEG biomarkers | 24 months
  P1, N1, P2, N2 and P3 waves, amplitudes and latencies - Elicitation of evoked potentials (ERP) will use the O-Kidia battery to elicit components associated with attention, stress, or anxiety
mobile EEG biomarkers | 24 months
  N170 waves, amplitudes and latencies as measures of episodic memory
mobile EEG biomarkers | 24 months
  Alpha-, theta, beta waves and their ratios as a measures of ADHD assessments.
UX/UI feasibility | 12 months
  Questionnaire (10-items) assessing the usability (UX/UI) for children, on a five-point likert type scale ranging 0 to 50 points, higher scores meaning better outcome.
Test-retrests for the O-Games battery | 24 months
  Significant changes of either or both scores at T2 compared with baseline (repeated testing), higher scores meaning better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Douet Vannucci, PhD, Principal Investigator — O-Kidia
Locations (2):
- France (2):
  - Association la Busserine, Marseille, Provence Alpes Cotes d'Azur
  - O-Kidia, Gardanne, Provence-Alpes-Côte d'Azur Region

REFERENCES:
- See also: O-Kida website — https://www.o-kidia.com